CLINICAL TRIAL: NCT05714800
Title: Endocardial Mapping of Left Atrium for Evaluation of Concomitant Surgical Ablation Lesions for Treatment of Atrial Fibrillation
Brief Title: Endocardial Mapping of Left Atrium for Evaluation of Concomitant Surgical Ablation Lesions
Acronym: PLAN-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, Electrophysiology specialist, University Medical Centre Ljubljana
Other Study IDs: PLAN-AF
Record Dates: First submitted 2023-01-22; First posted 2023-02-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: concomitant ablation; heart surgery; remapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Concomitant ablation is an effective treatment for patients with various types of atrial fibrillation undergoing heart surgery.

However, recurrences of tachycardias after concomitant ablation can happen and seem to be mostly related to reentry mechanism resulting in atrial tachycardias.

The aim of the study is to perform invasive re-mapping of ablated regions in the atria to assess durability of ablation lesions and prevalence of conduction gaps that can be targets for additional ablation to lower longterm arrhythmia recurrence.

DETAILED DESCRIPTION:
Patients after concomitant ablation for treatment of atrial fibrillation will be enrolled. At ablation procedure pulmonary veins will be isolated and additional ablation lines will be performed in the left atrium (posterior wall box lesion, connecting lesion to the mitral annulus, connecting lesion to the left atrial appendage,...) and the right atrium (intercaval connecting lesion, cavotricuspid isthmus lesion,...) and left atrial appendage will be excluded (suture and excision, clipping device,...) at the discretion and expertise of the operator. Radiofrequency and/or cryoablation will be used at the discretion and expertise of the operator.

Invasive mapping with a high density mapping catheter connected to a three-dimensional electro-anatomical mapping system will be performed to assess pulmonary vein isolation and linear lesion durability 3 months after the initial concomitant ablation. Potential gaps will be identified and ablated with a radiofrequency ablation catheter.

Participants will be followed-up clinically and with holter ECG before and after the invasive re-mapping procedure up to the first year after the concomitant ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for any kind of elective heart surgery having also indication (EHRA and/or HRS guidelines) to undergo concomitant ablation for any type of atrial fibrillation

Exclusion Criteria:

* life expectancy of less than one year,
* severe heart failure with left ventricular ejection fraction below 35%,
* emergency surgery due to a life threatening condition such as acute aortic dissection, papillary muscle rupture, acute endocarditis, major trauma,...

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery for treatment of heart valve disease, surgical coronary artery revascularization, benign cardiac tumors,... having also any type of atrial fibrillation with an indication to undergo concomitant ablation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-06-03 (Estimated); Study Completion 2025-06-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of conduction gaps | 3 months
  Prevalence of conduction gaps in pulmonary vein isolation lines and linear ablation lines found at the invasive re-mapping procedure
Prevalence of atrial fibrillation/tachycardia before and after delayed invasive re-mapping | 12 months
  ECG and holter ECG will be performed before and after the re-mapping procedure to assess possible change in prevalence related to closure of potential conduction gaps at the re-mapping procedure

CONTACTS AND LOCATIONS:
Overall Officials: Matevž Jan, MD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lippi G, Sanchis-Gomar F, Cervellin G. Global epidemiology of atrial fibrillation: An increasing epidemic and public health challenge. Int J Stroke. 2021 Feb;16(2):217-221. doi: 10.1177/1747493019897870. Epub 2020 Jan 19. PMID 31955707
- [Background] Kornej J, Borschel CS, Benjamin EJ, Schnabel RB. Epidemiology of Atrial Fibrillation in the 21st Century: Novel Methods and New Insights. Circ Res. 2020 Jun 19;127(1):4-20. doi: 10.1161/CIRCRESAHA.120.316340. Epub 2020 Jun 18. PMID 32716709
- [Background] Badhwar V, Rankin JS, Damiano RJ Jr, Gillinov AM, Bakaeen FG, Edgerton JR, Philpott JM, McCarthy PM, Bolling SF, Roberts HG, Thourani VH, Suri RM, Shemin RJ, Firestone S, Ad N. The Society of Thoracic Surgeons 2017 Clinical Practice Guidelines for the Surgical Treatment of Atrial Fibrillation. Ann Thorac Surg. 2017 Jan;103(1):329-341. doi: 10.1016/j.athoracsur.2016.10.076. PMID 28007240
- [Result] McClure GR, Belley-Cote EP, Jaffer IH, Dvirnik N, An KR, Fortin G, Spence J, Healey J, Singal RK, Whitlock RP. Surgical ablation of atrial fibrillation: a systematic review and meta-analysis of randomized controlled trials. Europace. 2018 Sep 1;20(9):1442-1450. doi: 10.1093/europace/eux336. PMID 29186407
- [Result] McCarthy PM, Kruse J, Shalli S, Ilkhanoff L, Goldberger JJ, Kadish AH, Arora R, Lee R. Where does atrial fibrillation surgery fail? Implications for increasing effectiveness of ablation. J Thorac Cardiovasc Surg. 2010 Apr;139(4):860-7. doi: 10.1016/j.jtcvs.2009.12.038. PMID 20304134